CLINICAL TRIAL: NCT05864508
Title: Interest of Oxytocin as an Adjuvant Treatment of Psycho-educational Measures in Challenging Behaviors in Children With Autism Spectrum Disorders and Moderate to Severe Intellectual Disability: Feasibility and Safety Study.
Acronym: OT-DEFI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0500; 2022-000254-28 (EudraCT Number)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum disorder; Oxytocin; Intellectual disability; Challenging behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intranasal oxytocin (Experimental): intranasal oxytocin treatment once a day during 6 weeks
  Interventions: Drug: Oxytocin nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — intranasal oxytocin treatment once a day during 6 weeks

SUMMARY:
The investigation team propose in this study to specifically evaluate the feasibility of using oxytocin in the form of an intranasal spray in a specific population of children with autism spectrum disorder and intellectual disability. The lack of studies centered on this population on the one hand, and on the other hand the severity of challenging behaviors presented by these children, make questionable the direct transfer of methods of care used in patients who do not present these challenging behavior. In this sense, the establishment of oxytocin treatment in these children requires a preliminary phase of feasibility assessment before being able to consider a comparative trial of the randomized clinical trial type.

DETAILED DESCRIPTION:
Taking into account:

* Intellectual disability comorbidity as a risk factor for challenging behaviors in the population with autism spectrum disorder;
* behavioral difficulties inherent in the presence of these behaviors, which are all potential obstacles to the administration of a treatment and therefore above all raise the question of the feasibility of administering such a treatment;
* the difficulty for children associating autism spectrum disorder of severe intensity and intellectual disability to benefit from clinical and paraclinical examinations given the concern generated by such examinations and challenging behaviors which can then occur in them, raising the question of feasibility monitoring protocol
* results of Oxytocin administration obtained in patients with autism spectrum disorder without associated intellectual disability;
* the favorable drug safety profile of oxytocin in children with autism spectrum disorder of the same age but without challenging behaviors;
* the extreme need for an effective treatment to control challenging behaviors in children with autism spectrum disorder with associated intellectual disability,

the investigation team propose in this study to specifically evaluate the feasibility of using oxytocin in the form of an intranasal spray in a specific population of children with autism spectrum disorder and intellectual disability. The lack of studies centered on this population on the one hand, and on the other hand the severity of challenging behaviors presented by these children, make questionable the direct transfer of methods of care used in patients who do not present these challenging behavior. In this sense, the establishment of oxytocin treatment in these children requires a preliminary phase of feasibility assessment before being able to consider a comparative trial of the randomized clinical trial type.

ELIGIBILITY:
Inclusion Criteria:

* Minor benefiting from a social security scheme.
* Diagnosis:autism spectrum disorder according to the Diagnostic and Statistical Manual DSM -5 of severe intensity;
* Comorbidities:
* Moderate to severe intellectual disability
* Presence of challenging behavior objectified by means of clinical examination and the ABC and ABC-I scales
* Multi-professional psycho-educational and re-educational care : global and coordinated interventions associating, according to the needs, educational interventions by targeted objectives, therapeutic interventions involving functions that do not develop spontaneously, adaptation of the environment by structuring time and space, in close collaboration with the families.
* If prescribed psychotropic treatments (antipsychotics, anxiolytics, hypnotics/sedatives, antidepressants, psychostimulants and antiepileptics), the dosages must be stable for 3 months*
* Understanding of French by both parents (if applicable) and ability for both parents to understand, in particular, the instructions for administering the product and to answer questionnaires.
* Informed consent signed by the holders of parental authority

Exclusion Criteria:

* The refusal of the holders of parental authority
* Pregnant girls, determined by a positive baseline blood pregnancy test
* Criteria respecting the Syntocinon SPC:

  * Hypersensitivity to Syntocinon
  * Hyponatremia < 135 mmol/L
  * Hypokalaemia < 3.5 mmol/L
  * Hypertension or hypotension
* Behavioral intolerance to the intranasal route
* Hepatic impairment (ALT and/or AST > 3N)
* Kidney failure (creatinine > 3 N)
* History of an ECG considered to be clinically significant abnormal (validated by a cardiologist)
* Type 1 or 2 diabetes
* Prolongation of the QT interval and/or family history of QT prolongation linked to an identified genetic etiology (QTc prolongation threshold > 460 ms). **
* History of epilepsy or seizures
* Sexually active women of childbearing age without effective contraception*
* Breastfeeding women
* Severe cardiovascular disease (tachycardia, bradycardia, arrhythmias, hypertension, hypotension, myocardial ischemia)
* Latex allergy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
percentage of children with complete OT administration protocol | Week 14
  percentage of children who will complete the OT administration protocol
percentage of children with complete monitoring protocol | week 14
  percentage of children who will complete the monitoring protocol

CONTACTS AND LOCATIONS:
Overall Officials: Julie ANDANSON, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No